CLINICAL TRIAL: NCT06142019
Title: Pulse Oximeter Accuracy in Healthy Humans During Hypoxia
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 21-35637
Record Dates: First submitted 2023-09-21; First posted 2023-11-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hypoxia; Skin Pigmentation
MeSH Terms: conditions — Hypoxia; Pigmentation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Controlled desaturation (hypoxemia) — Stable hypoxemia is created in healthy subjects by having them breathe hypoxic air mixtures

SUMMARY:
The aim of this project is to test the accuracy of pulse oximeters during mild, moderate and severe hypoxia. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxygen. This study will be done on healthy male or females between the age group of 18-50.

DETAILED DESCRIPTION:
This study is to determine the accuracy of pulse oximeters, which measure blood oxygen by shining light through fingers, ears or other parts of the body, without requiring blood sampling.

The aim of this project is to test the accuracy of pulse oximeters during mild, moderate and severe hypoxia. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a laboratory hemoximeter).The data obtained is submitted by pulse oximeter manufacturers to the FDA for device approval.

Studies normally involve 10-14 normal adult volunteer paid subjects, with 20-25 1-2 ml arterial blood samples from each subject obtained at different steady-state levels of hypoxia from 70-100%. Blood samples obtained from an arterial line are measured in a hemoximeter to determine true saturation value. Some sponsors may not require any blood sampling. Some sponsors may require additional blood samples, up to 35 samples may be drawn. Readings from the test pulse oximeters are recorded and compared to these "gold-standard" blood values. The pulse oximeter probes may be located at a variety of sites on the subjects, including fingers, toes, ears, forehead, scalp and bridge of the nose. These detector-probes are all non-invasive.

The level of hypoxia is measured and controlled by the investigator. A computer program that displays a prediction, breath by breath, the arterial oxygen saturation, (SaO2) of the study subject. SaO2 is computed from end-expired Po2 and Pco2 as determined by mass spectrometer gas analysis. This information permits the inspired gas mixture of air, plus CO2 and nitrogen, to be adjusted by an operator watching the value computed after each expiration on an analog meter. This computer-estimated saturation is adjusted by the operator to one of 6 levels of predicted saturation, and is held stable for about 30 seconds at each level. Two or three "runs" are conducted per subject. Each "run" lasts 10-15 min and 4 to 5 plateaus are tested per run. The manufacturer may choose the target values. Plateaus are typically sought at 96%, 87%, 77%, 92%, 82% and 72%. Other manufacturers have asked for an equal number of data points but with all points between 70% and 100%. Some sponsors may also request additional variables to be measured during testing including high or low CO2, where subjects will be asked to hyperventilate; low perfusion, where subjects will be asked to lay flat, or with their head up or down; testing pulse oximeters during motion, or with the subject's hand fixed to a motion machine. The subject's will be informed by the study staff and in the consent form if any of these additional procedures apply.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>35).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population consists of healthy volunteers between 18-50 years of age across all ethnic and racial backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
SpO2 | 08/01/2025
  Reading on pulse oximeter device which is an estimate of the patient's blood oxygen level.

SECONDARY OUTCOMES:
Blood gas SO2 | 08/01/2025
  Arterial blood gas sample results showing exact SpO2 levels. SpO2 ranges from 1% to 100%. Our target SpO2 levels are between 67% and 100%.
Skin Pigmentation by ITA | 08/01/2025
  ITA stands for individual typology angle from a spectrophotometer which is an objective measurement of skin pigmentation. The categories for the ITA scale are the following: > 55 Very Light, 41 to 55 Light, 28 to 41 Intermediate, 10 to 28 Tan, -30 to 10 Brown, < -30 Dark.
Finger Diameter | 08/01/2025
  Finger diameter is measured to ensure that the pulse oximeters being tested work with a variety of finger sizes. Finger diameter is measured in mm.
Skin Pigmentation by Monk Scale | 08/01/2025
  The Monk scale is a subjective categorization of skin pigmentation. The Monk Scale is a 10 shade scale designed to to be easy-to-use for development and evaluation of technology while presenting a more representative range of skin tones than other common qualitative scales. The Monk Scale is from A to J. A being the lightest skin color and J the darkest.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, MD, PhD, Principal Investigator — University of California at San Francisco
Locations (1):
- Hypoxia Lab, UCSF Department of Anesthesia and Perioperative Care, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feiner JR, Bickler PE, Mannheimer PD. Accuracy of methemoglobin detection by pulse CO-oximetry during hypoxia. Anesth Analg. 2010 Jul;111(1):143-8. doi: 10.1213/ANE.0b013e3181c91bb6. Epub 2009 Dec 10. PMID 20007731
- [Background] Feiner JR, Severinghaus JW, Bickler PE. Dark skin decreases the accuracy of pulse oximeters at low oxygen saturation: the effects of oximeter probe type and gender. Anesth Analg. 2007 Dec;105(6 Suppl):S18-S23. doi: 10.1213/01.ane.0000285988.35174.d9. PMID 18048893
- [Background] Bickler PE, Feiner JR, Severinghaus JW. Effects of skin pigmentation on pulse oximeter accuracy at low saturation. Anesthesiology. 2005 Apr;102(4):715-9. doi: 10.1097/00000542-200504000-00004. PMID 15791098